CLINICAL TRIAL: NCT00596947
Title: Randomized, Prospective Single-center Study Comparing a Rapid Discontinuation of Corticosteroids (Steroid Withdrawal) With Corticosteroid Therapy in Kidney Transplantation Using Mycophenolate Mofetil and Tacrolimus Maintenance Therapy
Brief Title: Prednisone Withdrawal Versus Prednisone Maintenance After Kidney Transplant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: due to low study enrollment
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Simin Goral, Director, Polycystic Kidney Disease Clinic, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 803242
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2011-03-21 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-03

CONDITIONS: Transplants and Implants
Keywords: kidney transplantation; tacrolimus; Prograf; mycophenolate mofetil; CellCept; corticosteroid withdrawal; prednisone withdrawal; prednisone maintenance; rabbit antithymocyte globulin; Thymoglobulin
MeSH Terms: interventions — Prednisone; Steroids; Methylprednisolone; Adrenal Cortex Hormones; thymoglobulin; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone Withdrawal (Experimental): Participants randomized to the prednisone withdrawal group, received 4 medications to prevent rejection. Thymoglobulin (rabbit antithymocyte globulin) was given intravenously in the operating room at the time of transplant. Subsequent intravenous doses were administered to participants an inpatient or outpatient for a total of 3 to 5 doses. Participants also began taking Prograf (tacrolimus) and CellCept (mycophenolate mofetil)orally within 24 hours of transplant and continued indefinitely. The steroids were initially given in the operating room intravenously at time of transplant as Solu-medrol (methylprednisolone)and were then switched to daily oral prednisone doses. The participant's dose of prednisone was rapidly decreased until it was completely eliminated by day 6 post-transplant.
  Interventions: Drug: prednisone; Drug: rabbit antithymocyte globulin; Drug: Tacrolimus; Drug: Mycophenolate mofetil
- Prednisone Maintenance (Active Comparator): Participants randomized to the prednisone maintenance group, received 4 medications to prevent rejection. Thymoglobulin (rabbit antithymocyte globulin) was initiated intravenously in the operating room at the time of transplant. Subsequent intravenous doses were administered an inpatient or outpatient for a total of 3 to 5 doses. Participants began taking Prograf (tacrolimus) and CellCept (mycophenolate mofetil)orally within 24 hours of transplant and continued on them indefinitely. The steroids were initially given intravenously in the operating room at time of transplant as Solu-medrol (methylprednisolone) and were then switched to daily oral prednisone tablets. Participants remained on all drugs according to their doctor's standard of care, and the prednisone was not be eliminated.
  Interventions: Drug: rabbit antithymocyte globulin; Drug: Tacrolimus; Drug: Prednisone; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: prednisone — In this group, participants had prednisone rapidly decreased until completely eliminated by day 6 after transplant. Participants began on 500mg of intravenous methylprednisolone on the day of transplant, followed by the following doses of oral prednisone: 160mg on day 1, 120mg on day 2, 80mg on day 3, 40mg on day 4, 20mg on day 5, none from day 6-on.
  Other Names: Deltasone; Steroids; Methylprednisolone; Corticosteroids
  Arms: Prednisone Withdrawal
Drug: rabbit antithymocyte globulin — Participants in both groups received 3 to 5 doses of an intravenous medication to prevent rejection called Thymoglobulin (rabbit antithymocyte globulin) as per our standard of care. This drug was dosed at 1.5 milligrams/killograms per dose and dosing was then based on body weight. The dose was decreased in half or held if the participant had a low white blood cell count or if the participant a low platelet count. The first dose was given intravenously in the operating room and subsequent intravenous doses were administered either while participants were inpatients or outpatients for a total of 3 to 5 doses for a total of up to 6mg/kg. The number of doses was based on transplant kidney function and risk factors for rejection.
  Other Names: RATG; Thymoglobulin; Polyclonal antibody
Drug: Tacrolimus — Participants in both groups received tacrolimus per our standard of care. This medication helped to prevent rejection and was initially dosed at 0.1-0.2 milligrams/killograms/day in two divided doses, given orally, based on participant's body weight. We then looked at the trough levels of this medication(the lowest level before the next dose), and aimed to keep the trough level between 5-10 nanograms/milliliter throughout the study.
  Other Names: Prograf
Drug: Prednisone — Participants in this group continued on prednisone indefinitely. Participants began with 500mg of intravenous methylprednisolone on the day of transplant, followed by the following doses of oral prednisone: 160mg on day 1, 120mg on day 2, 80mg on day 3, 40mg on day 4, 20 mg days 5-9, 15 mg day 10-19, 10 mg day 20-24, 7.5 mg day 25-29, and 5mg from day 30-on indefinitely.
  Other Names: Deltasone; Steroids; Methylprednisolone; Corticosteroids
  Arms: Prednisone Maintenance
Drug: Mycophenolate mofetil — Participants in both groups received mycophenolate mofetil by mouth twice daily indefinitely. Dosing for patients in the Prednisone withdrawal group was 1000mg orally twice daily. The dose was decreased or held at the discretion of the physician, for side effects such as low white blood cell count, or low platelet count, or if the participant experienced stomach side effects such as heartburn, nausea, vomiting or diarrhea.
  Other Names: mmf; CellCept
  Arms: Prednisone Withdrawal
Drug: Mycophenolate mofetil — Participants in both groups received mycophenolate mofetil by mouth twice daily indefinitely. Dosing for patients in the Prednisone maintenance group was 500 mg orally twice daily. The dose was decreased or held at the discretion of the physician, for side effects such as low white blood cell count, or low platelet count, or if the participant experienced stomach side effects such as heartburn, nausea, vomiting or diarrhea.
  Other Names: mmf; CellCept
  Arms: Prednisone Maintenance

SUMMARY:
The purpose of the study was to determine if rapid discontinuation of corticosteroids (also known as prednisone withdrawal) and maintenance immunosuppression with Prograf (tacrolimus) and CellCept (mycophenolate mofetil) while using Thymoglobulin (Rabbit antithymocyte globulin) will give similar safety and efficacy results compared to continuation of corticosteroids (also known as prednisone maintenance) and standard maintenance immunosuppression with Prograf (tacrolimus), CellCept (mycophenolate mofetil) while using Thymoglobulin (Rabbit antithymocyte globulin).

DETAILED DESCRIPTION:
Corticosteroids (one specific type is prednisone) have been used in clinical transplantation for more than 30 years. There are many side effects of corticosteroids including significant bone disease, diabetes (elevated blood sugar levels), fluid retention and hypertension (high blood pressure), psychosis, peptic ulcer disease, hyperlipidemia (elevated lipid levels such as cholesterol and triglycerides), obesity (overweight), acne, and susceptibility to infections. It is hoped that the new generation of potent immunosuppressive medications (such as Prograf and CellCept) will permit avoidance or withdrawal of corticosteroids for the majority of patients to avoid both short- and long-term complications of corticosteroid use in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* First time kidney transplant recipients who receives a kidney from a cadaveric, living related or living unrelated donor
* Age greater than 18 years and less than 75 years
* Caucasian recipients
* Patients with current low panel reactive antibody (PRA) levels (<10%)
* Patients with signed and dated informed consent
* Women of childbearing potential must have a negative pregnancy test at baseline and agree to use a medically acceptable method of contraception throughout the treatment period.

Exclusion Criteria:

* Other than Caucasian ethnicity
* Patients with HIV+ or
* Patients with HbsAg+ or Hepatitis C positive
* Patients with a history of malignancy in the past 5 years
* Patients with active systemic or localized major infection
* Patients with a history of chronic steroid use for other diseases

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simin Goral, MD, Principal Investigator — University of Pennsylvania-Renal Electrolyte and Hypertension Division
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was terminated early due to low enrollment.
Groups:
- Prednisone Withdrawal: Participants randomized to the prednisone withdrawal group , were started on 4 drugs; Thymoglobulin (Rabbit antithymocyte globulin) Prograf (tacrolimus), CellCept (mycophenolate mofetil) and corticosteroids initially given as Solu-medrol (methylprednisolone) through a vein in the arm, and then given orally daily as prednisone tablets. The dose of prednisone for participants in this group was rapidly decreased until it was completely eliminated by day 6 after transplant.
- Prednisone Maintenance: Participants randomized to the prednisone maintenance arm were started on 4 drugs; Thymoglobulin (Rabbit antithymocyte globulin) Prograf(tacrolimus), CellCept (mycophenolate mofetil) and corticosteroids, initially as Solu-medrol(methylprednisolone) given through the vein in the arm and then as daily oral prednisone tablets. Participants in this arm received all drugs according to their doctors' standard of care and the prednisone was not be eliminated.
Period: Overall Study
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Started | 9 | 9
Completed | 3 | 6
Not Completed | 6 | 3
Not completed — study halted due to low enrollment | 5 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12.3) | 50.6 (13.2) | 49.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 9 | 5 | 14
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Acute Rejection Episodes
Description: Acute rejection episodes would have been measured by the number of participants who underwent a kidney transplant biopsy, and had the results of the biopsy reported as acute rejection by the transplant pathologist. Biopsies were only performed if clinically indicated. The cumulative number of participants with recorded rejection episodes by 6 and 12 months post-transplant would have been reported.
Time Frame: 6 and 12 months post-transplant
Population: data not interpretable due to low patient enrollment
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: The Number of Participants With Treatment Failures
Description: This measure was defined as the percentage of participants that did not remain on initial therapy (ie were withdrawn from each arm of the trial)
Time Frame: 12 months
Population: Unable to interpret data due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Length of Hospital Stay After Transplant
Description: The length of the hospital stay would have assessed the number of days a participant was in the hospital after the kidney transplant was performed. This is calculated from date of admission to date of discharge.
Time Frame: 12 months
Population: unable to interpret results due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: The Number of Participants With Hospital Readmissions
Description: The number of readmissions during the study period for each participant would have been assessed, as well as the reason for readmissions.
Time Frame: 12 months
Population: Unable to interpret data due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: The Length of Stay Associated With Hospital Readmissions
Description: The time from admission to discharge for each readmission for patients readmitted in the first 12 months post-transplant.
Time Frame: 12 months
Population: Unable to interpret data due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Participant Renal Function as Measured by MDRD Formula
Description: The above methods focus on estimating or determining actual glomerular filtration rate (GFR) (or renal function) of the kidney transplant. The MDRD (Modification of Diet in Renal Disease) calculation includes age, sex and serum creatinine would have provided an estimate of GFR. This was to be performed at 3,6 and 12 months post-transplant.
Time Frame: 3, 6 and 12 months
Population: Unable to interpret data due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Participant Renal Function as Measured by 24 Hour Urine Collection
Description: Results would have been reported from patients undergoing 24 hour urine collections at 3 and 12 months post-transplant. This is a way to measure glomerular function rate (GFR) or renal function.
Time Frame: 3 and 12 months post-transplant
Population: Unable to interpret data due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: The Number of Participants With Graft Survival
Description: The number of participants who did not experience graft failure (defined as return to dialysis) at 6 and 12 months would have been reported.
Time Frame: 6 and 12 months
Population: data not interpretable due to low patient enrollment
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Participant Survival
Description: The number of participants alive at 6 and 12 months post-transplant would have been posted as a measure of patient survival.
Time Frame: 6 and 12 months
Population: data not interpretable due to low patient enrollment
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: The Number of Participants With the Need for Rabbit Antithymocyte Globulin to Treat Rejection Episodes.
Description: The incidence and severity of rejection episodes per participant would have been identified by kidney transplant biopsy results read by a transplant pathologist. Treatment of rejection episodes in each participant would have been determined by the treating transplant physician.
Time Frame: 12 months
Population: unable to interpret results due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: The Number of Participants With Leukopenia
Description: All participants would have been assessed for the presence at any time during the trial of: leukopenia (defined by lab results as a white count less than 3,000 cells/uL).
Time Frame: 12 months
Population: unable to interpret results due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: The Number of Participants With Infections
Description: Participants would have been monitored throughout the study for any infectious complications as confirmed by the principal investigator. Patients would have been monitored by urine cytology and blood polymerase chain reaction for BK virus at baseline, and months 3, 6 and 12 post-transplant.
Time Frame: 12 months
Population: Unable to interpret data due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: The Number of Participants With Malignancy
Description: Participants would have been monitored throughout the study with any reports of malignancy being confirmed by principal investigator.
Time Frame: 12 months
Population: Unable to interpret data due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: The Number of Participants With Hypertension
Description: The number of participants who developed hypertension defined as blood pressure greater than 140/90 throughout the first 12 months of the study.
Time Frame: 12 months
Population: unable to interpret results due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: The Number of Participants With Hyperlipidemia
Description: Fasting lipid profiles were to be performed at 3,6 and 12 months post-transplant. Definitions based on ATP III guidelines.
Time Frame: 12 months
Population: Unable to interpret data due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: The Number of Participants With Bone Disease
Description: Bone densitometry by Computed tomography of peripheral skeleton and DEXA scans were performed at baseline (within one month after transplant) Urine and blood samples to measure markers of bone turnover: Alkaline phosphatase, pyridinoline, serum 1-25 vit D 3 levels (calcitriol) and 25 hydroxy vit D (calcidiol) levels and serum osteocalcin levels were drawn at baseline, 3, 6, 12 and 24 months.
Time Frame: baseline (within 1 month post-transplant), 3, 6, 12 and 24 months
Population: unable to interpret results due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: The Number of Participants With Post Transplant Diabetes Mellitus
Description: Glucose tolerance test performed in non-diabetic participants only at pre transplant in living donor recipients and at baseline (within 1 mo after transplant) and 6 mo and 12 months. Blood test for hemoglobin A1C in non diabetic participants only: at baseline, 3, 6, and 12 months.
  Insulin and C peptide levels at baseline, 3,6 and 12 months in all participants.
Time Frame: pre-transplant in living donor recipients, baseline (within one month post-transplant) and at 3, 6 and 12 months
Population: unable to interpret results due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: The Number of Participants With Weight Gain
Description: Height, weight will be used to calculate change in BMI for all participants.
Time Frame: 12 months
Population: unable to interpret results due to low number of patients enrolled.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 24 months post-transplant
Description: Patients and their data were reviewed by the principal investigator at regular follow-up visits, hospital readmissions and study visits.
Arm/Group | Prednisone Withdrawal | Prednisone Maintenance
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/9 | 4/9
Other Adverse Events (participants affected / at risk) | 8/9 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone Withdrawal (N=9) | Prednisone Maintenance (N=9)
gangrene (Vascular disorders) | 0 (0) | 1 (2) — Gangrene of left toe, same patient had gangrene of right toe in past
lower extremity edema (Renal and urinary disorders) | 0 (0) | 1 (1)
shortness of breath (Cardiac disorders) | 0 (0) | 1 (1)
hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
cytomegalovirus (Infections and infestations) | 0 (0) | 1 (1)
post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — was Epstein Barr positive, involved tongue and brain lesions, was ongoing at end of follow-up
lymphocele (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — Both events occurred post kidney transplant
perinephric fluid collection (Surgical and medical procedures) | 1 (1) | 0 (0) — This subject also had a prior lymphocele
fever (General disorders) | 2 (2) | 0 (0) — One patient had fever with perinephric fluid collection. Gram negative rods reported from fluid but not further identified. Other patient with fever was thought to have urinary tract infection, though no bug was identified.
hyperglycemia (Endocrine disorders) | 1 (2) | 1 (1) — Neither patient was noted to be diabetic pre-transplant.
acute cellular rejection (Immune system disorders) | 1 (1) | 1 (1)
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
seizure (Nervous system disorders) | 1 (1) | 0 (0)
3 Vessel CABG (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone Withdrawal (N=9) | Prednisone Maintenance (N=9)
wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1) — no bug identified
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) — bug identified as serratia marcescens
fungal infection of toes (Infections and infestations) | 1 (1) | 1 (1)
lower extremity edema (Renal and urinary disorders) | 2 (3) | 2 (4)
fatigue (General disorders) | 0 (0) | 1 (1)
shortness of breath (Cardiac disorders) | 0 (0) | 1 (1)
lightheadedness (Cardiac disorders) | 0 (0) | 1 (1) — same patient also had shortness of breath
hypertension (Renal and urinary disorders) | 1 (1) | 1 (1)
pain in right calf (General disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 0 (0) | 1 (1) — patient lost to follow-up
hyperkalemia (Renal and urinary disorders) | 0 (0) | 2 (4)
increased serum creatinine (Renal and urinary disorders) | 0 (0) | 2 (2)
leukopenia (Blood and lymphatic system disorders) | 2 (5) | 3 (4)
recurrence of gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
increased tacrolimus trough level (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
hyperglycemia (Endocrine disorders) | 2 (2) | 2 (2)
hypophosphatemia (Renal and urinary disorders) | 0 (0) | 1 (1)
hand tremors related to tacrolimus therapy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
lymphocele (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — hospitalization was not required for any of these cases
reaccumulation of peritransplant fluid collection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (4) — one patient also presented with concurrent vomiting
seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
anemia (Renal and urinary disorders) | 2 (2) | 2 (2)
osteopenia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) — One patient presented with concurrent osteoporosis of femoral region
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — patient presented with concurrent diarrhea
osteoporosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — patient presented with concurrent osteopenia of lumbar area
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
increased hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
bronchitis (Infections and infestations) | 1 (1) | 0 (0)
blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
insomnia (General disorders) | 2 (2) | 0 (0)
hypokalemia (Renal and urinary disorders) | 1 (1) | 0 (0)
hypercalcemia (Renal and urinary disorders) | 2 (2) | 0 (0)
hypocalcemia (Renal and urinary disorders) | 1 (1) | 0 (0)
leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
headache every morning (General disorders) | 1 (1) | 0 (0)
nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to low enrollment. Therefore no results beyond basic results section are reported due to uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No